CLINICAL TRIAL: NCT01914224
Title: Research for the Effectiveness of Combined Dietary Education of Low Sodium and High Potassium Consumption
Brief Title: Combined Dietary Education of Low Sodium and High Potassium Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DongGuk University (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Professor, MD, PhD, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13162MFDS106
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Prehypertension; Hypertension
Keywords: Prehypertension; Hypertension; Sodium; Potassium; renin; aldosterone
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): dietary education of low sodium and high potassium consumption
  Interventions: Behavioral: dietary education of low sodium and high potassium consumption
- Group 2 (Active Comparator): dietary education of low sodium consumption only
  Interventions: Behavioral: dietary education of low sodium consumption only

INTERVENTIONS:
Behavioral: dietary education of low sodium and high potassium consumption
  Arms: Group 1
Behavioral: dietary education of low sodium consumption only
  Arms: Group 2

SUMMARY:
Reduction in sodium consumption is important approach in public health care. In general population, reduction of sodium intake can reduce the future development of hypertension and cardiovascular event. Meanwhile, enhancement of potassium consumption is also important to reduce blood pressure and cardiovascular events. We hypothesized that combined education of low sodium and high potassium consumption is more effective in reducing blood pressure compared to dietary education of low sodium consumption only.

The present survey study was designed to test the effectiveness of combined education of low sodium and high potassium consumption in blood pressure reduction and improvement of other variables.

ELIGIBILITY:
Inclusion Criteria:

1. Prehypertension: with a systolic pressure from 120 to 139 mm Hg or a diastolic pressure from 80 to 89 mm Hg
2. Stage 1 hypertension: with a systolic pressure from 140 to 159 mm Hg or a diastolic pressure from 90 to 99 mm Hg

Exclusion Criteria:

1. Urinary tract disease
2. Secondary hypertension
3. Previous history of unstable angina, heart failure, myocardial infarction, coronary revascularization, cerebrovascular disease within 12 months
4. Ventricular tachycardia, atrial fibrillation and flutter
5. Hypertrophic cardiomyopathy
6. Known chronic kidney disease: serum creatinine = or > 2.0 mg/dL
7. Hypokalemia (<3.5 mmol/L) or hyperkalemia (>5.5 mmol/L)
8. Type 1 diabetes mellitus
9. Poorly controlled diabetes mellitus (HbA1C = or > 9%)
10. Unable to collect 24 hour urine sample
11. Pregnancy
12. Alcoholics
13. Severe liver disease
14. Night workers
15. Mental retardation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
changes of 24-hour ambulatory systolic and diastolic blood pressure | 3 months
  Effectiveness of combined dietary education of low sodium and high potassium consumption on changes of 24-hour ambulatory systolic and diastolic blood pressure, compared to dietary education of low sodium consumption only.

SECONDARY OUTCOMES:
changes of 24-hour urine sodium and potassium excretion | 3 months
  Difference of changes of 24-hour urine sodium and potassium excretion by each dietary education
changes of renin and aldosterone | 3 months
  Difference in changes of renin and aldosterone by each dietary education

OTHER OUTCOMES:
Changes of renin and aldosterone | 3 months
  Changes of renin and aldosterone by low sodium consumption
Changes of pulse wave velocity | 3 months
  Changes of pulse wave velocity by low sodium consumption
Changes of left ventricular mass index | 3 months
  Changes of left ventricular mass index by low sodium consumption

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, MD, PhD, Principal Investigator — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea